CLINICAL TRIAL: NCT01671956
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Study Designed to Evaluate the Safety, Efficacy, Pharmacokinetic and Pharmacodynamic Profile of Bertilimumab in Patients With Active Moderate to Severe Ulcerative Colitis
Brief Title: Evaluation of Safety, Efficacy, Pharmacokinetic and Pharmacodynamic of Bertilimumab in Patients With Active Moderate to Severe Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Immune Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Immune/BRT/UC-01
Record Dates: First submitted 2012-08-09; First posted 2012-08-24 (Estimated); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis, Active Moderate; Ulcerative Colitis, Active Severe
Keywords: IBD; UC; Colitis; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bertilimumab (Experimental): Bertilimumab 10 mg/kg will be administered by IV infusion over 30 minutes
  Interventions: Biological: Bertilimumab
- Placebo (Placebo Comparator): Phosphate buffered saline (PBS) placebo will be administered by IV infusion over 30 minutes.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Bertilimumab — IV infusion over 30 minutes, at Day 0, Day 14 and Day 28
  Arms: Bertilimumab
Biological: Placebo — IV infusion over 30 minutes, at Day 0, Day 14 and Day 28
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled, parallel group multi-center study in adult participants with active moderate to severe UC.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 to 70 years of age inclusive.
2. Diagnosed with active moderate to severe UC per standard diagnostic criteria for a minimum of 3 months:

   * Mayo score of 6-12 (inclusive) at the Screening Visit
   * Endoscopic evidence of active mucosal disease, as assessed by flexible sigmoidoscopy, with an Endoscopic Finding Sub-score of ≥2 (assessed centrally)
   * Rectal Bleeding Sub-score of ≥1
   * Physician's Global Assessment (PGA) Sub-score of ≥2.
3. Levels of eotaxin-1 in biopsied colon tissue of ≥100 pg/mg protein.
4. Adequate cardiac, renal and hepatic function as determined by the Investigator and demonstrated by screening laboratory evaluations and physical examination results; these findings must all be within normal limits or judged not clinically significant by the Investigator.

Exclusion Criteria:

1. History of colonic or rectal surgery other than hemorrhoidal surgery or appendectomy.
2. Currently receiving total parenteral nutrition (TPN).
3. Positive Clostridium difficile toxin stool assay.
4. Tested positive for active/latent mycobacterium tuberculosis (TB) infection.
5. Pregnant or breast-feeding, or plan to become pregnant during the study.
6. Males who are young and childless or planning to have more children in the future.
7. Known hypersensitivity to bertilimumab or any of the drug excipients.
8. History of infection requiring administration of any IV antibiotic, antiviral or antifungal medication within 30 days of Screening or any oral anti-infective agent within 14 days of Screening.
9. Severe UC evidenced by the following signs of toxicity: heart rate >100 beats/min at rest, temperature >37.8°C, hemoglobin <10.0 g/dL.
10. Ulcerative proctitis, defined as disease limited to less than 15 cm from the anal verge.
11. Received a vaccine or other immunostimulator within 4 weeks prior to screening.
12. Use of >4.8 g mesalazine or equivalent within 2 weeks prior to the screening visit. Mesalazine ≤4.8 g is allowed if the dose during the 2 weeks prior to the screening visit was stable.
13. Use of systemic corticosteroids exceeding the equivalent of 20 mg/day of prednisone within four weeks prior to the screening visit (see Section 6.9.1).
14. Change in dose of immunosuppressive drugs (e.g., corticosteroids, 6-mercaptopurine [6-MP], azathioprine) within four weeks prior to the screening visit.
15. Use of TNF-blockers (e.g., infliximab or adalimumab) within 60 days of the screening visit.
16. Use of chronic non-steroidal anti-inflammatory (NSAID) therapy. Occasional use of NSAIDs or acetaminophen for headache, arthritis, myalgias, menstrual cramps, etc., or daily use of low dose (81-162 mg) aspirin for cardiovascular prophylaxis is allowed.
17. Patients diagnosed with:

    * Crohn's disease
    * Diverticulitis or diverticulosis
    * Indeterminate colitis (inability to distinguish between UC and Crohn's disease [as assessed by the Investigator])
    * Microscopic colitis (collagenous or lymphocytic colitis)
    * Ischemic or infectious colitis
    * Clostridium difficile colitis within 90 days of the screening visit
    * Parasitic disease within 90 days of the screening visit
    * Systemic fungal infection within 90 days of the screening visit.
18. History of positive serology of hepatitis B or C, or human immunodeficiency virus (HIV) infection.
19. Congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, organ transplantation).
20. Clinically significant abnormal laboratory test results, unless regarded by the Investigator as related to UC, including but not limited to:

    * Hemoglobin level <10.0 g/dL
    * White blood cell count < 3 x 103/µL
    * Lymphocyte count < 0.5 x 103/µL
    * Platelet count <100 x 103/µL or >1200 x 103/µL
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 the upper limit of normal (ULN)
    * Alkaline phosphatase >3 ULN
    * Serum creatinine >2 ULN.
21. Active abuse of alcohol or drugs.
22. Known malignancy or history of malignancy that could reduce life expectancy.
23. Any condition, which in the opinion of the Investigator, would place the patient at an unacceptable risk if participating in the study protocol.
24. Participation in a clinical trial of an investigational (unapproved) product

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Research Site, Afula
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was initiated in Jul 2015 and was early terminated due to sponsor decision.
Groups:
- Bertilimumab: Participants with active moderate to severe ulcerative colitis received bertilimumab 10 mg/kg intravenous (IV) infusion biweekly for 12 weeks.
- Placebo: Participants with active moderate to severe ulcerative colitis received placebo IV infusion matched to bertilimumab biweekly for 12 weeks.
Period: Overall Study
Arm/Group | Bertilimumab | Placebo
Started | 20 | 12
Received at Least 1 Dose of Study Drug | 20 | 12
Completed | 18 | 10
Not Completed | 2 | 2
Not completed — Disease progression | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were exposed to any of the study treatments.
Groups:
- Bertilimumab: Participants with active moderate to severe ulcerative colitis received bertilimumab 10 mg/kg IV infusion biweekly for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Bertilimumab | Placebo | Total
Number analyzed (Participants) | 20 | 12 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 31
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity has not been collected.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 20 | 12 | 32
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Mayo Score at Day 56
Description: The Total Mayo score is an instrument designed to measure disease activity of ulcerative colitis and ranged from 0 (normal or inactive disease) to 12 (severe disease). It is a composite of 4 sub-scores: Stool frequency sub-score, rectal bleeding sub-score, endoscopic finding sub-score, and physician's global assessment sub-score, each of which ranges from 0 (normal) to 3 (severe disease). The sub-scores were summed to give a total score that ranged from 0-12. Change in mayo score was calculated as the sum of scores at Day 56 minus the sum of scores at Baseline divided by 14 for bertilimumab arm and sum of scores at Day 56 minus the sum of scores at Baseline divided by 6 for placebo arm.
Time Frame: Baseline, Day 56
Population: The modified intent to treat (mITT) analysis set included all randomized participants who received at least one dose of study treatment (placebo or bertilimumab) and had at least a full Mayo score at screening and at least one post-baseline partial Mayo score from visit 3 onwards. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Bertilimumab | Placebo
Number analyzed (Participants) | 14 | 6
scores on a scale | 2.7 [0 to 8] | 2.5 [1 to 6]

2. Secondary Outcome: Change From Baseline in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) Score at Day 56
Description: The UCEIS is the validated index for the assessment of overall endoscopic activity. The model incorporated the vascular pattern score (0-2), the presence of bleeding score (0-3) and the presence of erosions and ulcers score (0-3). The total score ranged from 0-8. Higher scores indicated more severe disease. Change in mayo score was calculated as the sum of scores at Day 56 minus the sum of scores at Baseline divided by 15 for bertilimumab arm and sum of scores at Day 56 minus the sum of scores at Baseline divided by 6 for placebo arm.
Time Frame: Baseline, Day 56
Population: The mITT analysis set included all randomized participants who received at least one dose of study treatment (placebo or bertilimumab) and had at least a full Mayo score at screening and at least one post-baseline partial Mayo score from visit 3 onwards. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bertilimumab | Placebo
Number analyzed (Participants) | 15 | 6
score on a scale | 1.2 [-3 to 5] | 0.4 [-1 to 2]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 90
Description: The safety analysis set included all participants who were exposed to any of the study treatments.
Arm/Group | Bertilimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/12
Other Adverse Events (participants affected / at risk) | 14/20 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bertilimumab (N=20) | Placebo (N=12)
Hypersenstivity (Immune system disorders) | 1 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bertilimumab (N=20) | Placebo (N=12)
Dysgeusia (Nervous system disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Ovulation pain (Reproductive system and breast disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study conducted by Immune Pharmaceuticals Inc. and was acquired by Alexion Pharmaceuticals, Inc after study completion, database lock, and report generation. Study was terminated early due to sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT01671956/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT01671956/SAP_001.pdf